CLINICAL TRIAL: NCT06160986
Title: Multidisciplinary Intervention for Adults With Chronic Graft Versus Host Disease
Brief Title: Horizons Chronic Graft-Versus-Host-Disease Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Lara Traeger, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230656
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Graft Vs Host Disease; Coping Skills; Quality of Life; Stem Cell Transplant Complications
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Horizons Group (Experimental): Participants will receive the Horizons Group intervention for up to 8 weeks.
  Interventions: Behavioral: Horizons Group Intervention

INTERVENTIONS:
Behavioral: Horizons Group Intervention — The Horizons Group intervention in English or Spanish language (per participant preference) contains 8 weekly group sessions delivered via video conference by a bone marrow transplant clinician and behavioral health specialist, over approximately 8 weeks, approximately 1.5 hours per session every week. The intervention pairs state-of-the-science information about survivorship and chronic graft versus host disease with self-management strategies. Intervention sessions will be delivered via video conference (Zoom), which participants may access by computer, laptop, tablet, or smart phone. As part of the intervention, participants will have access to an intervention manual and audio-recorded relaxation exercises to support learning and skills practice.

SUMMARY:
This research is being done to evaluate the feasibility of the Horizons Program, a group-based behavioral intervention, to enhance quality of life in patients with chronic graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

* underwent allogeneic hematopoietic stem cell transplant
* have moderate to severe chronic graft versus host disease
* currently receiving care at the Sylvester Comprehensive Cancer Center Bone Marrow Transplant Program
* able to participate in a group intervention in English or Spanish language

Exclusion Criteria:

* comorbid conditions or cognitive impairment that the treating clinician believes prohibits informed consent or participation in the intervention
* vulnerable patients, defined here as prisoners and pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participant enrollment | Baseline (pre-intervention) to 10-week follow-up
  Participant enrollment will be demonstrated if ≥50% eligible participants enroll
Percentage of participant attendance | Baseline (pre-intervention) to 10-week follow-up
  Participant attendance will be demonstrated if ≥80% participants complete ≥4 of 8 sessions
Percentage of participant retention | Baseline (pre-intervention) to 10-week follow-up
  Participant retention will be demonstrated if ≥80% participants are retained in the study at week 10.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No